CLINICAL TRIAL: NCT03969407
Title: Determination of the Best Positive End-expiratory Pressure (PEEP) Based on Oxygenation or Driving Pressure in Patients With Acute Respiratory Distress Syndrome After Cardiac Thoracic Surgery
Brief Title: Determination of the Best Positive End-expiratory Pressure (PEEP)
Acronym: DROP
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01760-55
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-05

CONDITIONS: Positive Expiratory Pressure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of the best positive end-expiratory pressure (PEEP) based on oxygenation or driving pressure in patients with acute respiratory distress syndrome (ARDS) after cardiothoracic surgery

The use of a positive end-expiratory pressure in acute respiratory distress syndrome is obvious in ARDS management. On the one hand it serves to fight against the reduction of functional residual capacity (FRC) and enable the limitation of hypoxia; and on the other hand it allows the limitation of "opening/closing" lesions in pulmonary alveoli which lead to increase "bio trauma".

However elevated PEEP has harmful effect such as hemodynamic effect on the right ventricle and distension on healthy part of the lung.Other adverse effects are: decreasing cardiac output, increased risk of barotrauma, and the interference with assessment of hemodynamic pressures.

Ideally the adjustment of PEEP level must be done by taking into account each patient characteristic. PEEP titration based on blood gas analysis is one of the most used techniques by physicians.

Current guidelines for lung-protective ventilation in patients with acute respiratory distress syndrome (ARDS) suggest the use of low tidal volumes (Vt), set according to ideal body weight (IBW) of the patient, and higher levels of positive end-expiratory pressure (PEEP) to limit ventilator-induced lung injury (VILI). However, recent studies have shown that ARDS patients who are ventilated according to these guidelines may still be exposed to forces that can induce or aggravate lung injury.

Driving pressure (DP) is the difference between the airway pressure at the end of inspiration (plateau pressure, Ppl) and PEEP.

Driving pressure may be a valuable tool to set PEEP. Independent of the strategy used to titrate PEEP, changes in PEEP levels should consider the impact on driving pressure, besides other variables such as gas exchange and hemodynamics. A decrease in driving pressure after increasing PEEP will necessarily reflect recruitment and a decrease in cyclic strain. On the contrary, an increase in driving pressure will suggest a non-recruitable lung, in which overdistension prevails over recruitment.

The main purposes of this study are to assess the optimal PEEP based on the best driving pressure or the best oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* All Patients admitted for intensive care with acute respiratory distress syndrome intubated according to the criteria of the Berlin Consensus

Exclusion Criteria:

* Undrained pneumothoraces
* Hemodynamic instability defined by increased need of vasopressors and / or an systolic arterial pressure below 90 mmHg
* Hypovolemic shock
* Bronchopleural fistula
* High intracranial pressure

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient admitted to adult intensive care with ARDS following cardiothoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Best PEEP level based on the best driving pressure value | 1 DAY
Best PEEP level based on the best oxygenation value defined by the PaO2/FiO2 ratio. | 1 DAY

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No